CLINICAL TRIAL: NCT01157338
Title: Clinical Significance of Retinal Emboli During Diagnostic and Therapeutic Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Dr Javad Kojuri, Shiraz University of medical sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1123
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Cardiac Catheterization; Retina; Embolism
Keywords: Catheter; coronary artery disease; embolus; stroke; retinal emboli
MeSH Terms: conditions — Embolism; Coronary Artery Disease; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diagnostic cardiac catheterization (Active Comparator): patients with diagnostic cardiac catheterization
  Interventions: Procedure: diagnostic cardiac catheterization
- therapeutic cardiac catheterization (Active Comparator): patient with angioplasty
  Interventions: Procedure: therapeutic cardiac catheterization

INTERVENTIONS:
Procedure: diagnostic cardiac catheterization — coronary intervention: angiography
  Arms: diagnostic cardiac catheterization
Procedure: therapeutic cardiac catheterization — cardiac catheterization: angioplasty
  Arms: therapeutic cardiac catheterization

SUMMARY:
Retinal emboli is a common phenomenon in cardiac catheterization. In this study the investigators evaluate the incidence of retinal emboli post diagnostic and therapeutic cardiac catheterization over 300 patients. The incidence was 6.3% and had no clinical sequel on visual acuity and visual field.

DETAILED DESCRIPTION:
Background and Purpose Cardiac catheterization may cause retinal embolization, a risk factor for cerebrovascular emboli and stroke. We describe the incidence of clinically silent and apparent retinal emboli following diagnostic and interventional coronary catheterization and associated risk factors.

Methods Three hundred selected patients attending a tertiary referral center for diagnostic and therapeutic cardiac catheterization were studied. Direct retinal examination and examination of the visual field and acuity were done before and after catheterization by a retinal specialist.

ELIGIBILITY:
Inclusion Criteria:

* every patient with diagnostic and therapeutic cardiac catheterization

Exclusion Criteria:

* patient refusal to follow up ophthalmology
* abscence of coronary disease in angiogram
* abnormal retinal angiogram prior to study

Ages: 52 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
retinal emboli
  retinal emboli detected by retinal especialist by direct examination

SECONDARY OUTCOMES:
visual field
  visual field detected by ophthalmologist
visual acuity
  snellen chart by ophthalmologist

CONTACTS AND LOCATIONS:
Locations (1):
- shiraz University of medical sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kojuri J, Mehdizadeh M, Rostami H, Shahidian D. Clinical significance of retinal emboli during diagnostic and therapeutic cardiac catheterization in patients with coronary artery disease. BMC Cardiovasc Disord. 2011 Jan 21;11:5. doi: 10.1186/1471-2261-11-5. PMID 21255443